CLINICAL TRIAL: NCT01846871
Title: A Phase II Study of Tivozanib in Recurrent Glioblastoma
Brief Title: Tivozanib for Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Elizabeth R. Gerstner, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-069
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tivozanib (Experimental): 1.5 mg daily for 3 weeks, with 1 week off.
  Interventions: Drug: Tivozanib

INTERVENTIONS:
Drug: Tivozanib
  Other Names: AV-951

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the study drug tivozanib is still being studied. It also means that the FDA has not yet approved tivozanib for your type of cancer.

Tivozanib is an anti-angiogenesis medicine that fights different types of cancer by blocking the blood supply to the tumor, so that the tumor does not receive the nutrients it requires to grow.

In this research study, we are looking to see what effects, good and bad, tivozanib will have on you and your disease.

DETAILED DESCRIPTION:
If you are willing to participate in this study, you will be asked to undergo some screening tests and procedures that confirm you are eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out taht you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. The screening process may include the following: a medical history, mini-mental status exam, physical exam, performance status, electrocardiogram, blood tests, urine test. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

If you take part in this research study, you will be given a study drug-dosing calendar for each treatment cycle. Each treatment cycle lasts 28 days (4 weeks) during which time you will be taking the study drug once daily for 3 weeks and then no study drug for the last week of each cycle. The diary will also include special instructions for taking the study drug.

During all cycles you will have a physical exam and you will be asked questions about your general health and specific questions about any problems that you might be having and any medications you may be taking.

Standard contrast-enhanced (CE) MRI scans will be done prior to all odd-numbered study cycles. Vascular MRI scans will be done prior to start of treatment, Day 1 of treatment and prior to all even-numbered cycles. These studies will be done in the Charlestown Navy Yard.

We would like to keep track of your medical condition for up to 24 months after your last dose of study treatment. We would like to do this by calling you on the telephone once a year to see how you are doing. Keeping in touch with you and checking your condition every year helps us look at the long-term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma that has progressed based on imaging or surgery
* Measurable disease
* No more than 3 prior chemotherapy regimens
* Must have recovered from toxicity of prior therapy. An interval of at least 3 months must have elapsed since the completion of the most recent course of radiotherapy; at least 3 weeks since last non-nitrosourea containing chemotherapy regimen or molecularly targeted agent; at least 6 weeks since the completion of a nitrosourea containing chemotherapy regimen
* Life expectancy of at least 12 weeks
* Able to tolerate MRIs
* Willing to use adequate, highly effective contraception measures while on study and for at least 45 days after the last dose of study drug

Exclusion Criteria:

* Pregnant or breastfeeding
* Major surgical procedure or significant traumatic injury within 28 days of starting therapy; or minor surgical procedure within 7 days
* Receiving other study agents
* Prior therapy with an anti-VEGF agent
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tivozanib
* Receiving any medications or substances that are inhibitors or inducers of CYP450 enzymes
* Significant cardiovascular disease
* Non-healing wound, bone fracture or skin ulcer
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis or other gastrointestinal condition with increased risk of perforation; abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug
* Uncontrolled intercurrent illness
* Significant thromboembolic or vascular disorders within 6 months prior to administration of first dose of study drug
* Significant bleeding disorders within 6 months prior to administration of first dose of study drug
* Currently active second primary malignancy
* HIV positive and on combination antiretroviral therapy
* Inability to swallow capsules, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of study drugs, major resection of the stomach or small bowel, or gastric bypass procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gerstner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tivozanib: 1.5 mg daily for 3 weeks, with 1 week off.
  Tivozanib
Period: Overall Study
Arm/Group | Tivozanib
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tivozanib
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 62 [51 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive and Progression Free After 6 Months
Description: To determine the number of patients with recurrent glioblastoma (GBM) alive and progression free 6 months (PFR6) after start of tivozanib therapy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tivozanib
Number analyzed (Participants) | 10
Participants | 1

2. Secondary Outcome: Number of Participants With Treatment Related Serious Adverse Events
Description: The number of participants with serious adverse events deemed possibly, probably, or definitely related to treatment. Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).
Time Frame: From the start of treatment until disease progression, unacceptable toxicity, or death; median duration of approximately 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tivozanib
Number analyzed (Participants) | 10
Participants | 0

3. Secondary Outcome: Median Overall Survival
Description: Overall survival is measured from the start of treatment until the time of death.
Time Frame: From the start of treatment until the time of death, median duration of approximately 8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tivozanib
Number analyzed (Participants) | 10
Months | 8.1 [5.2 to 12.5]

4. Secondary Outcome: Median Progression-Free Survival
Description: Progression free survival is measured as the amount of time from the start of treatment until the time of death or disease progression. Progressive disease was assessed using MacDonald Criteria
  Progressive disease: Progressive neurologic abnormalities not explained by causes unrelated to tumor 40 progression (example: anti-epileptic drug or corticosteroid toxicity, electrolyte abnormalities, hyperglycemia, etc.) or a greater than 25% increase in the volume of the tumor by MRI scan. If neurologic status deteriorates on a stable or increasing dose of corticosteroids, or if new lesions appear on serial MRI scans, this will also be considered PD.
Time Frame: From the start of treatment until death or progression, median duration of approximately 2 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tivozanib
Number analyzed (Participants) | 10
Months | 2.3 [1.5 to 4]

5. Secondary Outcome: Best RANO Criteria Response
Description: Best response as assessed by Response Assessment in Neuro-Oncology (RANO) criteria.
  Complete response
  * disappearance of all enhancing disease
  * sustained for at least 4 weeks
  * stable/improved non-enhancing FLAIR/T2W lesions
  * no new lesions
  * no corticosteroids
  * clinically stable/improved
  Partial response >50% or more decrease of all measurable enhancing lesions
  * sustained for at least 4 weeks
  * no progression of non-measurable disease
  * stable/improved non-enhancing FLAIR/T2W lesions
  * no new lesions
  * stable/reduced corticosteroids
  * clinically stable/improved
  Stable disease
  * does not qualify for complete response, partial response or progression
  * stable non-enhancing FLAIR/T2W lesions
  * stable or reduced corticosteroids
  * clinically stable
  Progression >25% or more increase in enhancing lesions despite stable/increasing steroid dose
  * increase in non-enhancing FLAIR/T2W lesions, not attributable to other non-tumor causes
  * any new lesion
  * Clinical deterioration
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Tivozanib
Number analyzed (Participants) | 10
Participants
  Complete response | 1
  Partial response | 1
  Stable disease | 4
  Progressive disease | 4

6. Secondary Outcome: Steroid Dosage
Description: The number of participants on steroids at baseline and the number of participants that increased or decreased their use of steroids during the course of treatment. Participants that required an increase and decrease in steroid use over the course of treatment were counted in both categories.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Tivozanib
Number analyzed (Participants) | 10
participants
  On steroids at baseline | 4
  Decreased dosage | 3
  Increased dosage | 4
  No change | 4

7. Secondary Outcome: Change in Tumor Volume
Description: Change in volume of the tumor in cubic centimeters at the given time points as compared to baseline
Time Frame: Baseline, Cycle 1 day 2, pre-cycle 2, pre-cycle 3 (1 cycle= 4 weeks)
Population: Measurements were not available for all participants at pre-cycle 2 and pre-cycle 3
Measure: Median (Inter-Quartile Range); unit: Cubic Centimeters
Groups:
- Tivozanib (Baseline): 1.5 mg daily for 3 weeks, with 1 week off.
  Tivozanib
- Tivozanib (Cycle 1 Day 2); Tivozanib (Pre-cycle 2); Tivozanib (Pre-cycle 3): 1.5 mg daily for 3 weeks, with 1 week off.
Arm/Group | Tivozanib (Baseline) | Tivozanib (Cycle 1 Day 2) | Tivozanib (Pre-cycle 2) | Tivozanib (Pre-cycle 3)
Number analyzed (Participants) | 10 | 10 | 9 | 8
Cubic Centimeters | 17.37 [5.18 to 31.11] | -2.012 [-6.08 to -0.79] | -2.75 [-5.68 to 3.19] | -3.53 [-18.28 to 1.76]
Statistical Analysis 1: Comparison: Tivozanib (Pre-cycle 3); Test type: Other; p = 0.70, t-test, 2 sided

8. Secondary Outcome: Median Apparent Diffusion Coefficient (ADC)
Description: Change in the the median ADC value from baseline at the given timepoints. Apparent diffusion coefficient (ADC) is a measure of the magnitude of diffusion (of water molecules) within tissue.
Time Frame: Baseline, Cycle 1 day 2, pre-cycle 2, pre-cycle 3 (1 cycle= 4 weeks)
Measure: Median (Inter-Quartile Range); unit: mm2/s
Arm/Group | Tivozanib (Baseline) | Tivozanib (Cycle 1 Day 2) | Tivozanib (Pre-cycle 2) | Tivozanib (Pre-cycle 3)
Number analyzed (Participants) | 10 | 10 | 10 | 10
mm2/s | 0.0013 [0.0011 to 0.0015] | -0.00009 [-0.00014 to -0.00005] | -0.00024 [-0.00032 to -0.00011] | -0.00023 [-0.0003 to -0.00004]
Statistical Analysis 1: Comparison: Tivozanib (Baseline) vs Tivozanib (Pre-cycle 3); Test type: Other; p = 0.028, t-test, 2 sided

9. Secondary Outcome: Median Ktrans
Description: Change in the the median Ktrans value from baseline at the given time points. The volume transfer constant (Ktrans) reflects the efflux rate of gadolinium contrast from blood plasma into the tissue extravascular extracellular space (EES)
Time Frame: Baseline, Cycle 1 day 2, pre-cycle 2, pre-cycle 3 (1 cycle= 4 weeks)
Measure: Median (Inter-Quartile Range); unit: mL/min/100 mL
Arm/Group | Tivozanib (Baseline) | Tivozanib (Cycle 1 Day 2) | Tivozanib (Pre-cycle 2) | Tivozanib (Pre-cycle 3)
Number analyzed (Participants) | 10 | 10 | 10 | 10
mL/min/100 mL | 0.032 [0.026 to 0.054] | -0.01468 [-0.025 to -0.010] | -0.024 [-0.032 to -0.022] | -0.030 [-0.045 to -0.022]
Statistical Analysis 1: Comparison: Tivozanib (Baseline) vs Tivozanib (Pre-cycle 3); Test type: Other; p = 0.0019, t-test, 2 sided

10. Secondary Outcome: Relative Oxygen Saturation
Description: The change in relative O2 saturation from baseline to the given time points. Oxygen saturation is a relative measure of the concentration of oxygen that is dissolved or carried in a given medium as a proportion of the maximal concentration that can be dissolved in that medium.
Time Frame: Baseline, Cycle 1 day 2, pre-cycle 2, pre-cycle 3 (1 cycle= 4 weeks)
Population: One participants was not available for assessment for the cycle 1 day 2 measurement
Measure: Median (Inter-Quartile Range); unit: proportion of possible O2 concentration
Arm/Group | Tivozanib (Baseline) | Tivozanib (Cycle 1 Day 2) | Tivozanib (Pre-cycle 2) | Tivozanib (Pre-cycle 3)
Number analyzed (Participants) | 10 | 9 | 10 | 10
proportion of possible O2 concentration | 0.64 [0.55 to 0.68] | -0.057 [-0.11 to -0.00003] | -0.0041 [-0.060 to 0.063] | -0.097 [-0.12 to -0.017]
Statistical Analysis 1: Comparison: Tivozanib (Baseline) vs Tivozanib (Pre-cycle 3); Test type: Other; p = 0.033, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the start of treatment until disease progression, unacceptable toxicity, or death; median duration of approximately 2 months.
Arm/Group | Tivozanib
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tivozanib (N=10)
Seizure (Nervous system disorders) | 2 (2)
Edema cerebral (Nervous system disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tivozanib (N=10)
Abducens nerve disorder (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Ear and labyrinth disorders - Other, cerumen in right ear (Ear and labyrinth disorders) | 1 (1)
Ear and labyrinth disorders - Other, hearing loss in right ear (Ear and labyrinth disorders) | 1 (1)
Ear and labyrinth disorders - Other, Intermittent hearing loss (Ear and labyrinth disorders) | 1 (1)
Eye disorders - Other, Hemanopsia (Eye disorders) | 1 (1)
Eye disorders - Other, Retro Orbital pressure (Eye disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Gait disturbance (General disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (8)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Investigations - Other, SGOT elevated (Investigations) | 1 (1)
Investigations - Other, SGPT elevated (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Nervous system disorders - Other, Altered Coordination (right) (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, Cognitive Dysfunction (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, numbness right limbs (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, Speech impairment (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 4 (4)
Skin infection (Infections and infestations) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes